CLINICAL TRIAL: NCT00681551
Title: Intra-individual Comparison Study of Intravenously Administered Magnevist (SH L 451A) on Lesion Detection Ability in MRI After an Initial Dose of 0.1 mmol/kg and After an Additional Dose of 0.1 mmol/kg in Patients With Metastatic Brain Tumor
Brief Title: Magnevist (SH L 451A) Intra-individual Dose Comparison Study in Patients With Brain Metastasis
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Bayer (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Diagnostic
Other Study IDs: 91103; 305624
Record Dates: First submitted 2008-04-01; First posted 2008-05-21 (Estimated); Last update posted 2014-12-15 (Estimated); Status verified 2014-12

CONDITIONS: Brain Neoplasms
Keywords: Detection of brain metastasis by MRI; Magnevist; Brain metastasis; Meglumine gadopentetate
MeSH Terms: conditions — Brain Neoplasms | interventions — Gadolinium DTPA

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Arm 1 (Active Comparator)
  Interventions: Drug: Magnevist (SH L 451A)
- Arm 2 (Experimental)
  Interventions: Drug: Magnevist (SH L 451A)

INTERVENTIONS:
Drug: Magnevist (SH L 451A) — Magnevist at a dose of 0.1 mmol/kg
  Arms: Arm 1
Drug: Magnevist (SH L 451A) — Magnevist at a dose of 0.1 mmol/kg and another 0.1 mmol/kg 30minutes later.
  Arms: Arm 2

SUMMARY:
To verify the number of metastatic brain tumors detected in contrast-enhanced MRI, which is the primary variable, increases after an additional dose of Magnevist (SH L 451A) comparing images after an initial dose (0.1 mmol/kg) with those after an additional dose (0.1 mmol/kg, a total dose of 0.2 mmol/kg) intra-individually in patients with metastatic brain tumors. Safety was also to be assessed.

ELIGIBILITY:
Inclusion Criteria:

* Patients who are confirmed to have 1-5 metastatic brain tumor by the latest contrast-enhanced cerebral CT or contrast-enhanced cerebral MRI, and the lesion(s) have not been treated by surgery or by stereotactic radiosurgery.

Exclusion Criteria:

* Patients who are scheduled to receive another contrast medium for MRI (except for oral agents) or iodine contrast medium (except for oral agents), or to undergo surgical procedures during the period from the day before administration of Magnevist (SH L 451A) to examination of safety on the following day.
* Patients who underwent or are scheduled to undergo radiotherapy during the period from 14 days before administration of Magnevist (SH L 451A) to examination of safety on the following day.
* Patients who were treated or are scheduled to be treated with anti-cancer agents (except for treatment only by the oral agents of the fixed dose continuously from 28 days or more before administration of Magnevist (SH L 451A)) during the period from 28 days before administration of Magnevist (SH L 451A) to examination of safety on the following day.

Min Age: 20 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 45 (Actual)
Dates: Start 2003-02; Study Completion 2004-03 (Actual)

PRIMARY OUTCOMES:
Diagnostic ability | MRI image in blinded read

SECONDARY OUTCOMES:
Visibility | MRI image in blinded read
Diagnostic confidence | MRI image in blinded read

CONTACTS AND LOCATIONS:
Overall Officials: Bayer Study Director, Study Director — Bayer
Locations (8):
- Japan (8):
  - Yokohama, Kanagawa
  - Osaka, Osaka
  - Hamamatsu, Shizuoka
  - Bunkyo-ku, Tokyo
  - Ōta-ku, Tokyo
  - Shinagawa-ku, Tokyo
  - Shinjuku-ku, Tokyo
  - Nakakoma-gun, Yamanashi